CLINICAL TRIAL: NCT00756782
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of TAC-101 in Combination With Transcatheter Arterial Chemoembolization (TACE) Versus TACE Alone in Asian Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of TAC-101 in Combination With TACE Versus TACE Alone in Asian Patients With Advanced Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to safety concerns.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAC101-204
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — TAC 101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients will receive TAC-101 20 mg (2 x 10-mg formulated tablets) administered orally every day with approximately 8 oz. water within 1 hour following a morning meal for 14 days followed by a 7-day recovery period, repeated every 21 days
  Interventions: Drug: TAC-101
- B (Placebo Comparator): Patients will receive placebo (two matching tablets) at same frequency and duration of active treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAC-101 — Patients will receive TAC-101 20 mg (2 x 10-mg formulated tablets) administered orally every day with approximately 8 oz. water within 1 hour following a morning meal for 14 days followed by a 7-day recovery period, repeated every 21 days.
  Arms: A
Drug: Placebo — Patients will receive placebo (two matching tablets) at same frequency and duration of active treatment
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TAC-101 after Transcatheter Arterial Chemoembolization (TACE) in patients with advanced, unresectable hepatocellular carcinoma (HCC) who are being scheduled for TACE.

DETAILED DESCRIPTION:
Transcatheter arterial chemoembolization (TACE) is a commonly performed procedure in the treatment of unresectable liver tumors for selected patients. TACE is a major palliative treatment for these patients. Most patients will have intrahepatic recurrence of their tumors following TACE. In this study, which will be conducted in Asian countries excluding Japan, TAC-101 will be administered as maintenance therapy after TACE compared with placebo therapy after TACE to patients with advanced HCC who are being scheduled for TACE and who either have not had any previous TACE procedures or who received their most recent TACE at least 120 days before signing the Informed Consent Form (ICF) and the TACE procedure resulted in complete necrosis, to determine if TAC-101 will enhance the benefits of TACE.

ELIGIBILITY:
Inclusion Criteria:

-A patient must meet all of the following inclusion criteria to be eligible for enrollment in this study and before undergoing the first TACE procedure of this study:

1. Has an HCC diagnosis by histology (can not have a mixed tumor type such as HCC and cholangiocarcinoma) OR by the following non-invasive criteria observed either within 14 days prior to first TACE or in the past.

   * One imaging technique (CT scan or magnetic resonance imaging [MRI] both with unenhanced plus hepatic arterial phase and portal venous phases) showing characteristic features in a focal lesion > 20 mm with arterial vascularization, or
   * Two dynamic imaging techniques (CT scan, MRI with unenhanced plus hepatic arterial phase and portal venous phases) showing characteristic features coincidentally in a focal lesion 10-20 mm with arterial vascularization.
2. Is TACE naïve or has received the most recent TACE procedure, which showed complete necrosis after treatment, at least 120 days before signing ICF.
3. Eligible to receive TACE and being scheduled to receive TACE.
4. Is ≥ 18 years of age.
5. Is not amenable to treatment with curative surgery, transplant, or percutaneous ablation, including RFA, percutaneous ethanol injection therapy (PEIT) and percutaneous microwave coagulation therapy (PMCT).
6. Have at least 1 measurable lesion that is ≥10 mm in size. Measurable lesions must be confirmed nodular type (not including only infiltration type) which demonstrated substantial hypervascularity by CT scan or MRI both with unenhanced plus hepatic arterial phase and portal venous phases. All measurable lesions must be targeted by the first TACE in this study

   * If there are ≥ 4 intrahepatic lesions, at least 1 must be ≥10 mm and all lesions must be <100 mm.
   * If there are < 4 intrahepatic lesions, at least one must be ≥ 30 mm and all lesions must be <100 mm.
   * No vascular invasion in main trunk and first order branch of portal vein or other large vessels (hepatic vein or inferior vena cava).
   * No extrahepatic tumor spread
7. Absence of extrahepatic abdominal tumors must be confirmed.
8. Has adequate organ function as defined by the following criteria:

   * White blood cell (WBC) count > 3,000/mm3
   * Platelet count > 60,000/mm3
   * Hemoglobin > 8.0 grams (g)/deciliter (dL)
   * Aspartate transaminase (AST) < 5 x ULN
   * Alanine transaminase (ALT) < 5 x ULN
   * Total bilirubin < 2.0 mg/dL
   * Albumin > 2.8 g/dL
   * Serum creatinine < 1.5 mg/dL
   * International normalized ratio (INR) ≤ 2.0
   * Triglyceride ≤ 2.5 x ULN.
9. Has a Child-Pugh classification of ≤ 8.
10. Has a Cancer of the Liver Italian Program (CLIP)68 score of 0, 1, 2 or 3.
11. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
12. Is willing and able to comply with schedule visits, treatment plans, laboratory tests, and other study procedures.
13. Provides written informed consent prior to the implementation of any study assessment or procedures.

Exclusion Criteria:

- Patients will be excluded from participation in the study if any of the following conditions are observed before undergoing the first TACE procedure:

1. Has only infiltration type of HCC.
2. Has extrahepatic metastasis of HCC including regional lymph node metastases.
3. Has had systemic chemotherapy (eg, sorafenib, doxorubicin), immunotherapy, or biologic therapy or radiotherapy for HCC, or treatment with TAC-101.
4. Received treatment with any of the following within the specified time frame:

   * Any major surgical procedure within 28 days prior to signing the ICF
   * Any red blood cell or thrombocyte transfusion, treatment with blood component preparation, albumin preparation, Granulocyte-Colony Stimulating Factor (G-CSF), or erythropoietin within 14 days prior to signing the ICF
   * Any intra-arterial chemotherapy (transcatheter injection) using lipiodol for HCC performed within 119 days prior to signing ICF.
   * Any local therapy such as alcohol injection, radiofrequency/ultrasound ablation, intraarterial chemotherapy (transcatheter arterial injection) for HCC performed within 28 days prior to signing the ICF
   * Any investigational agent within 28 days prior to signing the ICF
5. Has ascites, pleural effusions or pericardial fluid refractory to diuretic therapy.
6. Has clinical symptoms of hepatic encephalopathy.
7. Has active or uncontrolled clinically serious infection excluding chronic hepatitis.
8. Has a history of gastrointestinal (GI) bleeding in last 3 months.
9. Has previous or concurrent malignancy except for in situ carcinoma of the cervix, or other solid tumor treated curatively and without evidence of recurrence for at least 3 years prior to the study.
10. Has uncontrolled metabolic disorders or other nonmalignant organ or systemic diseases or secondary effects of cancer that induce a high medical risk and/or make assessment of survival uncertain.
11. Has any history during the last 3 years of deep vein thrombosis (DVT), pulmonary embolism (PE), myocardial infarction (MI), cerebrovascular accident (CVA), transient ischemic attack (TIA), unstable angina pectoris, or any other significant thromboembolic event (TE).
12. Has ejection fraction (EF) by echocardiogram (ECHO) or multi-gate acquisition (MUGA) that is outside of the normal range according to the site's institutional standard.
13. Has GI disease resulting in an inability to take oral medication.
14. Has had a liver transplant.
15. Has known allergy or hypersensitivity to TAC-101, doxorubicin, epirubicin, other anthracyclines, anthracenediones or any of the components used in the study drug formulations.
16. Has known hypersensitivity to iodinated contrast medium.
17. Is receiving therapeutic regimens of anticoagulants. However, use of low dose anticoagulants for prophylactic care of indwelling venous access device and use of low dose aspirin for prophylaxis are permitted.
18. Is taking medication known or suspected to predispose patient to an increased risk of VTE (eg, oral contraceptives, hormone replacement therapy, megestrol acetate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
radiologically proven progression-free survival (PFS) | Tumor Imaging assessments will be conducted at screening/baseline within 14 days prior to first TACE; every 8 weeks during treatment within 14 days prior to first TACE and every 8 weeks during follow-up period within 14 days prior to first TACE.

SECONDARY OUTCOMES:
Overall survival (OS) | Survival status obtained every 8 weeks during imaging follow-up period, from first TACE, patients contacted every 12 weeks until death or for at least 3 yrs after randomization of the last patient.
Time to appearance of remote new lesions (TTNLr) | Tumor Imaging assessments will be conducted at screening/baseline within 14 days prior to first TACE; every 8 weeks during treatment within 14 days prior to first TACE and every 8 weeks during follow-up period within 14 days prior to first TACE.
Objective tumor response rate (ORR) according to RECIST criteria (CR + PR) | Tumor Imaging assessments will be conducted at screening/baseline within 14 days prior to first TACE; every 8 weeks during treatment within 14 days prior to first TACE and every 8 weeks during follow-up period within 14 days prior to first TACE.
Effects on the plasma levels of alpha-fetoprotein (AFP and AFP-L3) | Blood samples for AFP and AFP-L3assessment obtained at Screening/ Baseline; every 8 weeks after first TACE during the treatment period; at the end of the treatment period; and every 8 weeks (± 2 weeks) from first TACE during imaging f/up period.
Number of post-randomization TACE procedures | The number of post-randomization TACE procedures per patient in the double-blind treatment period patient will be counted every 8 weeks during treatment from first TACE.
The adverse event (AE) profile and tolerability of TAC-101 therapy with TACE versus placebo therapy with TACE | AEs will be reported from the time a patient signs ICF through the period of patient follow-up (30 days after the last dose of study medication).
The relationship between the PK of TAC-101 and its metabolites and safety and efficacy parameters, including hepatic function | Pharmacokinetic blood samples will be collected (optional) at 4 hours (± 1 hour), 8 hours (± 1 hour), and 24 hours (± 1 hour) post-dose on Day 1 of treatment Cycle 1. The 24-hour sample must be collected prior to dosing on Day 2.
The biological effects of TAC-101 on selected RAR-related factors and growth factor VEGF-A | Blood samples collected at Screening/Baseline; every 8 weeks (± 2 weeks) after first TACE during the treatment period; at the end of the treatment period; at the Safety Follow-up visit (30 days after the end of study treatment).
The relationship between tumor gene expression (mRNA expression) of co-activators and co-repressors and efficacy parameters | Tissue samples collected at Screening/Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Benedetti, MD, Study Director — Taiho Oncology, Inc.